CLINICAL TRIAL: NCT03252132
Title: Resistance Training in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IDNC-DD2-MUSCLE
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2; Polyneuropathy Diabetes; Diabetes Complications; Diabetic Peripheral Neuropathy; Muscle Weakness; Fall Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Diabetes Complications; Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: International, randomized controlled training trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week resistance training (Active Comparator)
  Interventions: Other: 12-week resistance training
- No training (No Intervention)

INTERVENTIONS:
Other: 12-week resistance training — Training will consist of a minimum of 5 supervised training sessions every 2 weeks and each session will be approximately 60 minutes in duration. Patients will be performing resistance training consisting of at least 3 exercises affecting the largest muscle groups of the body, training the most basic movement patterns that work the entire body as a coordinated system. Patients will train according to a linear progressive model with a slow increase in weight every training session focusing on the flexors, extensors of the ankle and knee and on flexors, extensors and abductors of the hip.
  Arms: 12-week resistance training

SUMMARY:
This is a population-based study of type 2 diabetes patients with and without neuropathy recruited from the Danish National Type 2 Diabetes cohort (DD2).

Diabetic patients with neuropathy may suffer from incapacitating symptoms such as pain, muscle weakness and impaired balance. Muscle weakness may cause reduced balance and postural instability increasing the risk of frequent falls and thereby increased morbidity and mortality. Thus, diabetic neuropathy is associated with significant disabilities having major impact on activities of daily living and quality of life.

The effects of resistance training on neuropathy symptoms, muscle strength and muscle structure in patients with and with diabetic neuropathy will be examined.

DETAILED DESCRIPTION:
Perspective: The studies will likely improve the understanding of diabetic neuropathy and the relation between risk of falls in patients with and without motor dysfunction. The results may enable new and more precise recommendations for exercise in diabetic patients with diabetic neuropathy. In addition, the results may lead to a better understanding of the mechanisms underlying the effects of training. The improvement of motor function may lead to improved gait stability, fewer fall injuries and better quality of life for type 2 diabetes patients, resulting in lower morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes

Exclusion Criteria:

* Neuropathy due to any other cause

  * BMI >40
  * Pacemaker
  * Comorbidity that contraindicates exercise
  * History of stroke with affection of the lower extremities
  * Ischemic heart disease
  * Any other neurological disease
  * Pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Intraepidermal nerve fiber density (IENFD) | Change from baseline IENFD at 12 weeks
  1-2 small biopsies of 3 mm will be performed before and after the 12-week training period to evaluate small nerve fiber function.
Muscle strength (isokinetic strength) | Change from baseline IENFD at 12 weeks
  Isokinetic dynamometry will be used to determine the maximal isokinetic strength of the flexors and extensors at the knee, hip and ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Snopek, MD, Principal Investigator — Danish Pain Research Center, Aarhus University
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan KS, Overgaard K, Tankisi H, Karlsson P, Devantier L, Gregersen S, Jensen TS, Finnerup NB, Pop-Busui R, Dalgas U, Andersen H. Effects of progressive resistance training in individuals with type 2 diabetic polyneuropathy: a randomised assessor-blinded controlled trial. Diabetologia. 2022 Apr;65(4):620-631. doi: 10.1007/s00125-021-05646-6. Epub 2022 Jan 19. PMID 35048156